CLINICAL TRIAL: NCT06304103
Title: An Efficacy and Safety Study of AND017 for the Treatment of Anemia Due to Lower Risk Myelodysplastic Syndromes (MDS)
Brief Title: A Study of Efficacy and Safety of AND017 in Patients with Myelodysplastic Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AND017-MDS-206
Record Dates: First submitted 2023-03-22; First posted 2024-03-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AND017 capsules 4 mg (Experimental)
  Interventions: Drug: AND017
- AND017 capsules 12 mg (Experimental)
  Interventions: Drug: AND017
- AND017 capsules 30 mg (Experimental)
  Interventions: Drug: AND017

INTERVENTIONS:
Drug: AND017 — Administer AND017 once per day (QD)

SUMMARY:
This is a Phase 2, multicenter, randomized, open-lable, dose ranging study to evaluate the efficacy and safety of AND017 for the treatment of anemia due to lower risk Myelodysplastic syndromes (MDS) in patients subjects who are Red blood cell (RBC) non-transfusion dependent (NTD) and low transfusion burden (LTB).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of primary myelodysplastic syndrome with a PISS-R grading of very low, low or intermediate risk and a bone marrow primitive cell count < 5%, the time frame for this grading assessment should be at least 12 weeks prior to the first dose
2. Non-5q(del)-associated myelodysplastic syndrome.
3. Two non-transfused hemoglobin ≥ 6.0 g/dL and < 10.0 g/dL, averaged over the screening period, at least one week and more apart, and with no more than 1.3 g/dL difference between the two Hb.
4. Non-transfused subjects (NTD cohort) defined as no red blood cell transfusion in the 16 weeks prior to randomization or low transfusion load subjects defined as 3-7 pRBC units transfused in the 16 weeks prior to randomization and at least two different time points (LTB-1 cohort) or 1-2 pRBC units transfused at one time point in the 16 weeks prior to randomization ( LTB-2 cohort) (except in the case of transfusion for treatment of other comorbidities such as blood loss, surgery, etc.);
5. Baseline EPO level ≤ 500 mU/mL
6. Platelets ≥ 30,000 /mm3 and absolute neutrophil count ≥ 800/mm3
7. Adequate liver function with:

   * Total bilirubin <2 x upper limit of normal (ULN) (subjects with Gilbert's syndrome, i.e., unconjugated hyperbilirubinemia, have a total bilirubin <3 x ULN)
   * Aspartate aminotransferase (AST) <3 x ULN
   * Alanine aminotransferase (ALT) <3×ULN

Exclusion Criteria:

1. Diagnosed of secondary myelodysplastic syndrome or concurrent anemia from a cause other than the primary myelodysplastic syndrome.
2. Significant myelofibrosis (fibrosis ≥ 2+).
3. Planned clearing chemotherapy or whole brain spinal cord radiotherapy during the study period.
4. Previous diagnosis of MDS IPSS-R high or very high risk.
5. Prior or planned hematopoietic stem cell transplant during the study period.
6. Received granulocyte colony-stimulating factor (G-CSF), or thrombopoietin, or thrombopoietin receptor agonist therapy within 8 weeks prior to the first dose;
7. Treatment with antithymocyte globulin, azacitidine, decitabine, cyclosporine, thalidomide, or lenalidomide within 12 weeks prior to the first dose.
8. The presence of active infection or inflammatory disease requiring systemic anti-infective therapy, including concomitant autoimmune disease with inflammatory symptoms (e.g., generalized erythema, ankylosing spondylitis, rheumatoid arthritis, psoriatic arthritis, dry syndrome, celiac disease, etc.)
9. Concurrent retinal neovascularization requiring treatment (diabetic proliferative retinopathy, age-related exudative macular degeneration, retinal vein occlusion, macular edema, etc.)
10. Inability to take oral medications, or a history of gastrectomy, concomitant gastroparesis, or other conditions that may have an impact on the absorption of gastrointestinal medications (excluding gastric polyps or colonic polypectomy)
11. Clinically significant bleeding (including transfusions required to treat bleeding or bleeding resulting in a decrease in hemoglobin ≥ 2 g/dL) within 4 weeks prior to the first dose, or a bleeding constitutional or bleeding risk that has not been medically or surgically corrected.
12. Uncontrolled hypertension (more than one-third of identifiable diastolic blood pressure values ≥ 100 mmHg and/or systolic blood pressure ≥ 160 mmHg at 16 weeks prior to and including screening testing)
13. Comorbid heart failure (New York Heart Association [NYHA] class III or higher)
14. Medical history of significant liver disease or active liver disease at screening assessment
15. Have been treated with any other hypoxia-inducing factor-prolyl hydroxylase inhibitor (HIF-PHI) in the 8 weeks prior to the first dose
16. Have been treated with an erythropoietic ESA within 8 weeks prior to the first dose
17. Have been treated with an androgenic anabolic steroid, testosterone enanthate or methandrostenolone within 8 weeks prior to the first dose
18. Have been treated with an iron chelator within 8 weeks prior to the first dose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of HI-E/RBC-TI responding subjects | From baseline to up to Week 25
  * NTD cohort: non-transfused Hb levels ≥1.5 g/dL relative to baseline* during any 8-week period from baseline to 24 weeks post-dose.
  * LTB-1 cohort: No transfusion during any 8-week period from baseline to 24 weeks post-dose.
  * LTB-2 cohort: No transfusions during any 8-week period from baseline to 24 weeks post-dose and untransfused Hb levels ≥1.5 g/dL.
    * Hb baseline is the average of the two lowest Hb over the 16 weeks prior to the first dose

SECONDARY OUTCOMES:
For changes in mean transfusion units throughout the treatment period compared to baseline (mean transfusion units 16 weeks prior to first dose) | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  For changes in mean transfusion units throughout the treatment period compared to baseline (mean transfusion units 16 weeks prior to first dose)
For LTB cohorts, the average time required to reach first transfusion independence throughout the treatment period | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  For LTB cohorts, the average time required to reach first transfusion independence throughout the treatment period
Levels of reticulocyte count at each visit and change from baseline | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  Levels of reticulocyte count at each visit and change from baseline
Levels of hematocrit at each visit and change from baseline | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  Levels of hematocrit at each visit and change from baseline
Levels of mean corpuscular volume at each visit and change from baseline | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  Levels of mean corpuscular volume at each visit and change from baseline
Levels of mean corpuscular hemoglobin at each visit and change from baseline | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  Levels of mean corpuscular hemoglobin at each visit and change from baseline
Mean level and change from baseline in non-transfused Hb at each visit throughout the treatment period and | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  Mean level and change from baseline in non-transfused Hb at each visit throughout the treatment period
Mean level and change from baseline in non-transfused Hb throughout the first 8 weeks of treatment | Baseline, Week 3, 5, 7, and 9
  Mean level and change from baseline in non-transfused Hb throughout the first 8 weeks of treatment
Percentage of visits in which non-transfused Hb was maintained in this range after reaching two consecutive increases of ≥1.5 g/dL and ≥1.0 g/dL from baseline, respectively, throughout the treatment period | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  Percentage of visits in which non-transfused Hb was maintained in this range after reaching two consecutive increases of ≥1.5 g/dL and ≥1.0 g/dL from baseline, respectively, throughout the treatment period
Mean time required after two consecutive increases in non-transfused Hb ≥1.5 g/dL and ≥1.0 g/dL from baseline, respectively, throughout the treatment period | Baseline, Week 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, and 25
  Mean time required after two consecutive increases in non-transfused Hb ≥1.5 g/dL and ≥1.0 g/dL from baseline, respectively, throughout the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Yusha Zhu, MD, PhD, Study Director — Kind Pharmaceuticals LLC

IPD SHARING:
Plan to Share IPD: No